CLINICAL TRIAL: NCT03106532
Title: A Multicenter, Randomized, Placebo-controlled, Double-blind, Dose-finding Phase 2 Clinical Trial to Evaluate the Efficacy in Reduction of Intraocular Pressure and Safety of PHP-201 in Patients With Normal Tension Glaucoma
Brief Title: Evaluation of PHP-201 Ophthalmic Solution in Patients With Normal Tension Glaucoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: pH Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHP-201-S203
Record Dates: First submitted 2017-03-30; First posted 2017-04-10 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Normal Tension Glaucoma
MeSH Terms: conditions — Low Tension Glaucoma | interventions — sovesudil; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PHP-201 0.25% ophthalmic solution (Experimental): PHP-201 0.25% ophthalmic solution, TID
  Interventions: Drug: PHP-201 0.25% ophthalmic solution
- PHP-201 0.5% ophthalmic solution (Experimental): PHP-201 0.5% ophthalmic solution, TID
  Interventions: Drug: PHP-201 0.5% ophthalmic solution
- Placebo ophthalmic solution (Placebo Comparator): Placebo ophthalmic solution, TID
  Interventions: Drug: Placebo ophthalmic solution

INTERVENTIONS:
Drug: PHP-201 0.25% ophthalmic solution — 3 drops daily, 28 days
  Other Names: PHP-201
  Arms: PHP-201 0.25% ophthalmic solution
Drug: PHP-201 0.5% ophthalmic solution — 3 drops daily, 28 days
  Other Names: PHP-201
  Arms: PHP-201 0.5% ophthalmic solution
Drug: Placebo ophthalmic solution — 3 drops daily, 28 days
  Other Names: PHP-201
  Arms: Placebo ophthalmic solution

SUMMARY:
Evaluation of the optimal dose for the efficacy in reduction of intraocular pressure and safety of PHP-201 ophthalmic solution in patients with normal tension glaucoma

DETAILED DESCRIPTION:
Data collection (electronic case report forms), Data dictionary (MedDRA)

ELIGIBILITY:
Inclusion Criteria:

* 19 years and older, female and male
* IOP ≤21 mmHg
* Subject showing open angle finding, glaucomatous optic nerve damage and visual field defects
* BCVA ≥+0.2

Exclusion Criteria:

* Subject with the disease and surgery history that are not eligible to participate (acute closed angle glaucoma, narrow angle glaucoma, advanced glaucomatous loss, ocular trauma, eye surgery or laser surgery, unstable angina, myocardial infarction, uncontrolled hypertension and diabetes, etc)
* Subject who can't discontinue contact lenses
* Subject who can't discontinue topical/systemic IOP lowering medication

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-02 (Actual)

PRIMARY OUTCOMES:
Mean diurnal IOP change | 4 weeks
  Mean diurnal IOP change from baseline at post-treatment time point of 4 weeks

SECONDARY OUTCOMES:
The number of patient with adverse events | 28 days
  The number of patient with adverse events including ocular adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided